CLINICAL TRIAL: NCT06253832
Title: Surgical Conservative Management of Placenta Accreta Disorders
Brief Title: Conservative Management of Placenta Accreta Spectrum
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tunis University (Other)
Collaborators: University Tunis El Manar (Other)
Responsible Party: Principal Investigator, Haithem Aloui, university hospital assistant, Tunis University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMNT PAS
Record Dates: First submitted 2024-02-02; First posted 2024-02-12 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Placenta Accreta; Post Partum Hemorrhage; Blood Loss Massive
Keywords: Placenta accreta; Conservative management; Uncontrolled hemorrhage
MeSH Terms: conditions — Placenta Accreta; Postpartum Hemorrhage | interventions — Hysterectomy

STUDY DESIGN:
Intervention Model Description: comparer le traitement conservateur chirurgical à l'hystérectomie dans le traitement du placenta accreta
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- conservative surgery (Experimental): resective-constructive surgery: the excision of the placenta and its attachment site on the myometrium. Subsequently, uterine reconstruction is undertaken.
  Interventions: Procedure: conservative surgery for placenta accreta spectrum
- hysterectomy 1 (Active Comparator): Standard hysterectomy is performed
  Interventions: Procedure: hysterectomy
- hysterectomy 2 (Active Comparator): Standard hysterectomy is performed
  Interventions: Procedure: hysterectomy

INTERVENTIONS:
Procedure: conservative surgery for placenta accreta spectrum — The surgical procedure involved a midline incision for the laparotomy approach. Dissection of the uterus from the posterior bladder wall extended down to the cervix, with coagulation of the vesicouterine vessels. Hysterotomy was executed in the upper segment, just above the area of myometrial invasion. Hemostasis of the lower uterus was achieved through either square compression sutures or ligation of the colpouterine vessels. A conservative approach to uterine surgery was considered viable only under conditions of stable hemodynamics and when at least 2 cm of healthy myometrium was visibly intact above the cervix. For cases involving conservative resection, all myometrium affected by invasion and the entire placenta were excised. Subsequently, the uterus was reconstructed using a continuous stitching technique.
  Arms: conservative surgery
Procedure: hysterectomy — hysterectomy for placenta accreta spectrum
  Arms: hysterectomy 1
Procedure: hysterectomy — hysterectomy for placenta accreta spectrum
  Arms: hysterectomy 2

SUMMARY:
The resective-constructive surgery, detailed in prior research by Palacios-Jaraquemada JM, involves excising the placenta and its attachment on the myometrium, with modifications including the systematic use of a double JJ probe, omitting arterial ligation, and prioritizing careful dissection and reconstruction.

A prospective single-center study conducted from January 4, 2020 to February 2, 2024, at the Tunisian maternity ward including cases of placenta accreta, increta and percreta. Data on the estimation of blood loss, complications, transfusions and intensive care admissions were recorded. Diagnosis of placenta accreta was based on imaging and histopathology. The blood loss calculation incorporates total blood volume and changes in hematocrit.

DETAILED DESCRIPTION:
The surgical procedure known as resective-constructive surgery involves the excision of the placenta and its attachment site on the myometrium. This method has been detailed in prior research by Palacios-Jaraquemada JM, upon which we have built with some modifications.

Our modifications include the systematic placement of a double JJ probe under spinal anesthesia, omitting the ligation of hypogastric arteries or uterine arteries. Cesarean sections are performed at 37 weeks of gestational age. We prioritize ligating newly formed blood vessels between the uterus and surrounding structures, carefully dissecting the bladder, performing hysterotomy, and meticulously removing the placenta and its insertion bed until reaching healthy tissues. Subsequently, uterine reconstruction is undertaken.

Placental boundaries are identified through extrauterine palpation, followed by a transverse hysterotomy. Intrauterine palpation delineates the inferior margins of the placenta, guiding the resection of the placental bed. Closure is achieved through hysterorrhaphy. The JJ probe is removed post-surgery, and hemostasis is ensured through the modified B-Lynch suturing technique.

The prospective single-center study spanned from January 4, 2020, to February 2, 2024, encompassing the maternity and neonatology center in Tunis.

Data pertaining to operative time, blood loss, operative complications (such as organ or vessel injury), and postoperative complications (both early and late) were documented. Additionally, the success of the technique, units of blood transfusion administered, and admissions to the intensive care unit (ICU) were meticulously recorded.

Suspicion of placenta accreta was initially raised through pelvic MRI and ultrasonography. PAS was confirmed in all enrolled patients based on clinical history, image analysis (including ultrasound, Doppler, and MRI), and histopathological confirmation.

Patients lacking an intrasurgical or histopathological diagnosis of PAS were excluded from the statistical analysis.

Proficiency in the surgical technique, incorporating specialized hemostasis and dissection maneuvers, was attained by senior obstetricians who participated in 5-7 surgeries before independently managing cases. This approach aimed to ensure the initial reproducibility of the methodology.

The calculation of blood loss took into consideration the total blood volume (TBV), pre-partum hematocrit, and post-partum hematocrit, using the following formulas :

* Total Calculated Blood Loss (in milliliters of red blood cells) = Total blood volume * Percentage of blood loss
* Total Blood Volume = 0.75 x {[height (in inches) x 50] + [weight (in pounds) x 25]}
* Percentage of Blood Loss = (pre-partum hematocrit - post-partum hematocrit) / pre-partum hematocrit.

This approach ensured accurate assessment of blood loss during the procedures.

Sample Size:

In determining the sample size for our study, we employed a statistical formula applicable in the context of comparing mean values across two distinct groups, namely the experimental and control groups. This calculation is rooted in the t-test for independent samples.

The process entails the following critical steps:

1. Establishing the Significance Level (Alpha): Set at 0.05 to ensure 95% confidence.
2. Selecting the Study's Power (1 - Beta): Predetermined at 90%.
3. Assessing the Standard Deviations of Both Groups: Derived from pilot study data.
4. Identifying the Minimum Clinically Significant Difference (Delta): This represents the smallest difference we aim to detect in our study.

Pilot Study:

Initially, a pilot study was conducted to ascertain the standard deviations of the two groups and to gain an insight into the expected minimum difference.

Main Study:

Post-pilot study, we estimated the sample size. The "conservative surgical treatment" group was compared with two "hysterectomy" groups, sharing similar characteristics.

Description of Surgical Technique:

Our team has developed illustrative photos of the surgical method used as well as videos.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing scheduled or emergency cesarean section for placenta accreta

Exclusion Criteria:

* No signs of Placenta Accreta Spectrum upon artificial delivery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female pregnant subject
Enrollment: 36 (Actual)
Dates: Start 2020-01-04 (Actual); Primary Completion 2022-08-17 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Estimated blood loss | peroperatively
  Blood spoliation during procedure
Hemoglobin variation | First 24 hours]
  The difference between the Baseline concentration of Hemoglobin and the lowest hemoglobin concentration noted during the procedure
Transfusion requirements | First 24 hours
  Number of red blood cells units transfused
Procedure duration | peroperatively
  Time needed to perform surgery from incision to skin closure
Intensive care transfer rate | first 24 hours
  Intensive care transfer following surgery for placenta accreta

SECONDARY OUTCOMES:
Length of stay in ICU | time from surgery up to 30 days postoperative
  duration of the stay in the ICU following surgery for placenta accreta
Clotting disorders | time from surgery up to 30 days postoperative
  Assessed by the incidence of Intravascular disseminated coagulopathy
Bladder wound | Time from surgery up to 30 days postoperative
  Incidence of accidental bladder damage
Digestive wound | Time from surgery up to 30 days postoperative
  Incidence of accidental digestive lesion

CONTACTS AND LOCATIONS:
Overall Officials: Ben Marzouk Maghrebi, Professor, Study Chair — Tunis University Manar
Locations (1):
- Haithem Aloui, Manouba, Tunis Governorate, Tunisia

IPD SHARING:
Plan to Share IPD: Undecided